CLINICAL TRIAL: NCT06779318
Title: A Real-World Study Comparing Maintenance Chemotherapy With Tegafur, Gimeracil, and Oteracil Potassium (S-1) Versus Follow-Up Observation After Adjuvant Therapy for Resected Pancreatic Cancer With High Risk of Recurrence/Metastasis (MSPAC-1)
Brief Title: Maintenance Chemotherapy With S-1 vs. Observation After Adjuvant Therapy for Resected Pancreatic Cancer With High Risk of Recurrence/Metastasis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Min Tu, Associate Chief Physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSPAC-1
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer; Postoperative Adjuvant Therapy; Maintenance Therapy
Keywords: Maintenance Therapy; S-1
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-1 Maintenance Therapy (Experimental): S-1 monotherapy
  Interventions: Drug: S-1
- Observation Only (No Intervention): Participants in this arm will undergo follow-up observation according to the trial protocol, without receiving any antineoplastic drugs for maintenance therapy.

INTERVENTIONS:
Drug: S-1 — Tegafur, Gimeracil, and Oteracil Potassium (S-1) 40-60 mg per dose, orally (p.o.), twice daily (BID), from Day 1 to Day 28, with a 6-week cycle, for a total of 8 cycles; or from Day 1 to Day 14, with a 3-week cycle, for a total of 16 cycles.
  Arms: S-1 Maintenance Therapy

SUMMARY:
The goal of this real-world study is to learn if maintenance chemotherapy with Tegafur, Gimeracil, and Oteracil Potassium (S-1) can improve disease-free survival (DFS) compared to follow-up observation in patients with resected pancreatic cancer at high risk of recurrence or metastasis after adjuvant therapy. The main questions it aims to answer are:

* Does maintenance therapy with S-1 improve disease-free survival (DFS) compared to follow-up observation after standard treatment for resected high-risk pancreatic cancer?
* Does S-1 maintenance therapy improve overall survival (OS), distant disease-free survival (DDFS), and local recurrence-free survival (LRFS) compared to observation?
* What are the safety and tolerability profiles of S-1 maintenance therapy compared to observation? Researchers will compare two groups: the S-1 maintenance therapy group and the observation-only group, to see if S-1 improves survival outcomes and safety.

Participants will:

* Receive maintenance chemotherapy with S-1 based on body surface area dosing or be assigned to the observation group without drug intervention.
* Undergo imaging evaluations every 12 weeks to monitor for disease recurrence or metastasis.
* Report side effects and any adverse events during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed pancreatic cancer (originating from the pancreatic ductal epithelium);
2. Meets one of the following conditions: Pathologically confirmed as moderately differentiated, moderately to poorly differentiated, or poorly differentiated; or pathologic staging as: T3N0M0, T1-3N1-2M0, T4N0-2M0; or one or more surgical margins are R1 resected (R0 resection if no tumor cells are found more than 1mm from the margin, otherwise R1 resection); or involvement of the portal vein and/or superior mesenteric vein resection; or pre-adjuvant chemotherapy CA19-9 > 90 U/mL; or pre-adjuvant chemotherapy ctDNA testing positive;
3. Completed standard treatment: Received radical resection, postoperative adjuvant therapy (including adjuvant chemotherapy based on gemcitabine or fluorouracil), and radiotherapy (if applicable);
4. Eligible for oral medication;
5. Age ≥18 and ≤75, male or female;
6. ECOG performance status: 0 to 2;
7. Normal function of major organs as per the following criteria within 14 days prior to starting treatment:① Neutrophil count ≥ 1.5×10^9/L;② Platelet count ≥ 75×10^9/L;③ Hemoglobin ≥ 9.0 g/dL;④ AST ≤ 2.5×UNL (upper normal limit) (if liver metastasis present, AST ≤ 5×UNL);⑤ ALT ≤ 2.5×UNL (if liver metastasis present, ALT ≤ 5×UNL);⑥ Total bilirubin ≤ 1.5×UNL;⑦ Creatinine clearance (calculated using the Cockcroft-Gault formula) > 60 mL/min or serum creatinine ≤ 1.5×UNL;
8. Women of childbearing potential must have used reliable contraception within 7 days prior to enrollment and have a negative pregnancy test, and must be willing to use appropriate contraception during the study and for 6 months after the last dose of the investigational drug. For men, they must be surgically sterile or agree to use appropriate contraception during the study and for 3 months after treatment;
9. Expected survival time ≥6 months;
10. Voluntary participation in the study, signed informed consent, and demonstrated good compliance and cooperation during follow-up.

Exclusion Criteria:

1. Pancreatic cancer originating from non-pancreatic ductal epithelium, including pancreatic neuroendocrine tumors, pancreatic acinar cell carcinoma, pancreatoblastoma, and solid-pseudopapillary tumor;
2. Incomplete macroscopic resection (R2 resection);
3. Presence of distant metastasis (including malignant ascites and pleural effusion, peritoneal metastasis) or locally recurrent pancreatic cancer;
4. CA19-9 > 180 U/mL within 21 days before enrollment;
5. Severe liver dysfunction (AST/ALT > 3.5 times the upper limit of normal, alkaline phosphatase > 6 times the upper limit of normal), with liver drainage;
6. Known peripheral neuropathy (CTCAE ≥ Grade 2);
7. Participation in another clinical trial of cytotoxic drugs, targeted therapies, immunotherapies, etc., within the past 4 weeks, or received systemic chemotherapy, radiotherapy, or biological therapy within the past 4 weeks;
8. Concurrent or metachronous cancers with disease-free survival ≥ 5 years (excluding pancreatic cancer), except for cancers that have been cured or can be potentially cured with local excision (e.g., esophageal cancer, gastric cancer, colorectal cancer, cervical cancer, non-melanoma skin cancer, bladder cancer);
9. Factors that significantly affect oral drug absorption, such as difficulty swallowing, chronic diarrhea, or gastrointestinal obstruction; uncontrolled Crohn's disease or ulcerative colitis;
10. Clinically symptomatic serous effusions (including pleural effusion, ascites, pericardial effusion) requiring symptomatic treatment;
11. Pregnant or breastfeeding women; patients of childbearing potential unwilling or unable to take effective contraceptive measures;
12. Known allergy to the investigational drug, the class of the investigational drug, or its components;
13. Need for systemic corticosteroid treatment (except for local steroid pre-treatment);
14. History of interstitial lung disease (including interstitial pneumonia, pulmonary fibrosis, etc.) or CT findings of interstitial lung disease;
15. Active local or systemic infection requiring treatment;
16. Heart failure NYHA classification ≥ II or severe heart disease;
17. Known HIV infection or history of acquired immunodeficiency syndrome (AIDS) or active hepatitis B or C;
18. Toxicity not recovered (CTCAE > Grade 1) or previous anticancer surgery not fully recovered;
19. Patients deemed unsuitable for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | Up to 3 years
  Disease-Free Survival (DFS) is defined as the time from enrollment to the first occurrence of disease recurrence or death from any cause, whichever occurs first. If no recurrence occurs during the study, DFS is defined as the time from enrollment to the last confirmed date of disease-free status. For participants who withdraw from the study for reasons other than recurrence (e.g., initiation of other treatments), DFS will be censored at the time of withdrawal or the start of other treatment. For participants who are not censored, pre-planned sensitivity analyses will be conducted based on radiologically confirmed recurrence or death. New primary tumors will not be considered as recurrence events. The confirmed recurrence date will be the date of imaging showing relapse. If recurrence is confirmed through other clinical methods, the date of diagnosis will be used.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Overall Survival (OS) is defined as the time from enrollment to death from any cause. For participants who are alive at the last follow-up, OS will be censored at the last known date of survival. In cases of participants lost to follow-up, OS will be censored at the last date they were confirmed to be alive.
Distant Disease-Free Survival (DDFS) | Up to 3 years
  Distant Disease-Free Survival (DDFS) is defined as the time from enrollment to the first occurrence of distant metastasis or death from any cause, whichever occurs first. If no distant metastasis occurs, DDFS will be defined as the time from enrollment to the last confirmed date of no distant metastasis.
Local Recurrence-Free Survival (LRFS) | Up to 3 years
  Local Recurrence-Free Survival (LRFS) is defined as the time from enrollment to the first occurrence of local recurrence or death from any cause, whichever occurs first. If no local recurrence occurs, LRFS will be defined as the time from enrollment to the last confirmed date of no local recurrence.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Up to 3 years
  This outcome will assess the number of participants who experience treatment-related adverse events, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. These events will be monitored and categorized based on severity, with a focus on the relationship to the study treatment.
Quality of Life (QoL) | Up to 3 years
  Quality of Life will be measured using the EORTC QLQ-C30 (version 3), a widely used instrument to assess the health-related quality of life of cancer patients. The scores will be analyzed to evaluate changes in the quality of life during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China